CLINICAL TRIAL: NCT05116592
Title: Post Prostatectomy Incontinence After Enucleation Surgery
Brief Title: The Risk Factor and Outcome of Transient Incontinence After Prostate Enucleation Surgery
Acronym: PPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202003023RINA
Record Dates: First submitted 2021-10-13; First posted 2021-11-11 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2022-10

CONDITIONS: Benign Prostatic Hyperplasia; Incontinence
Keywords: transient incontinence,TURP
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Lower urinary tract symptoms caused by benign prostatic hyperplasia (BPH) are the most common urological problem among men. monopolar transurethral resection of the prostate (TURP), in which the enlarged prostate tissue is resected piece by piece using a monopolar electrode, has been the gold standard since the 1970s. It can substantially improve the maximal flow rate (Qmax), urinary symptoms (International Prostate Symptom Score, IPSS), and health-related quality of life (QOL), with long-term efficacy compared to medications or other minimally invasive treatments.4 5 However, monopolar TURP is a risky procedure because of the likelihood of severe complications such as massive bleeding or transurethral resection (TUR) syndrome.6 Therefore, it is of paramount importance to develop minimally invasive surgical techniques with outcomes similar to those of monopolar TURP, but with fewer side effects. Therefore, new energy system with different surgical methods developed after 2000s. Among all, Enucleation methods was proved to have better Qmax and IPSS after surgery than vaporization and resection methods. However, the risk of short-term transient incontinence was higher in enucleation than in resection methods.

Hence modified methods such as upside down, apical preservation methods, defining the limits of dissection proximal to external sphincter prior to enucleation of prostate were developed in order to reduce transient incontinence. Besides, the necessity of preoperative urodynamic study and biofeedback training, investigate the risk factors of transient incontinence are important issues. The study using prospective cohort design recruit 300 BPH patient receiving enucleation methods. To investigate the risk factors of transient incontinence and establish model to predict the incontinence. Besides we will evaluate different surgical methods and treatment methods to improve transient incontinence and the long-term results of different enucleation methods.

DETAILED DESCRIPTION:
Lower urinary tract symptoms caused by benign prostatic hyperplasia (BPH) are the most common urological problem among men. Approximately one-third of men over the age of 50 are affected by this problem. Surgical intervention is the most effective treatment for BPH, with around 100,000 procedures carried out annually in the United States. Of all surgical treatments, monopolar transurethral resection of the prostate (TURP), in which the enlarged prostate tissue is resected piece by piece using a monopolar electrode, has been the gold standard since the 1970s. It can substantially improve the maximal flow rate (Qmax), urinary symptoms (International Prostate Symptom Score, IPSS), and health-related quality of life (QOL), with long-term efficacy compared to medications or other minimally invasive treatments. However, monopolar TURP is a risky procedure because of the likelihood of severe complications such as massive bleeding or transurethral resection (TUR) syndrome. Therefore, it is of paramount importance to develop minimally invasive surgical techniques with outcomes similar to those of monopolar TURP, but with fewer side effects.

Since the 2000s, new energy systems for BPH surgical interventions quickly became popular, including systems that use bipolar energy and various laser systems, such as the holmium laser, potassium-titanyl-phosphate (KTP) laser, thulium laser, and diode laser. The trend in BPH surgical therapy has shifted from monopolar TURP to laser therapies and bipolar TURP over the past 10 years. Bipolar energy can be used to incise, resect, and vaporize prostate tissue using different electrodes. Holmium and thulium laser beams are mainly absorbed by water and act as incisional lasers. The KTP laser is selectively absorbed by hemoglobin and debulks prostate tissue through vaporization. The diode laser is absorbed by water and hemoglobin can therefore vaporize and incise prostate tissue. These new methods all use normal saline instead of distilled water to avoid hyponatremia. They can be further divided into three types according to their treatment principles: resection methods (resection of prostate tissue piece by piece), vaporization methods (vaporization of excessive prostate tissue), and enucleation methods (peeling the enlarged prostate from the prostate capsule).

Enucleation methods was proved to have better Qmax and IPSS after surgery than vaporization and resection methods. In a network meta-analysis, enucleation methods, including bipolar enucleation of prostate , holmium, thulium, and diode laser enucleation of prostate, yielded greater Qmax values at 6-12-months after surgery than did the resection and vaporization methods, and the difference could still be observed at 24-36 months after treatment. The advantages of the enucleation over vaporization methods were mainly observed in large prostates. Enucleation methods also achieved better IPSS than resection and vaporization methods, although the difference was not statistically significant. The new methods were generally safer than monopolar TURP. They were less likely to require patient transfusion, cause blood clot tamponade, lead to postoperative hemoglobin decline, or cause TUR syndrome.

However, the risk of short-term transient incontinence was higher in enucleation than in resection methods. Compared with resection methods, enucleation methods had more events of short-term transient urinary incontinence than resection methods. (odds ratio (OR)=1.91, 95% Confidence interval (CI); 1.35 to 2.71) Liu et al compared bipolar enucleation with bipolar TURP and found that after Foley removal, the incontinence rate was higher in enucleation than in resection at 24 hours (35.6 % vs 18.9%, p<0.01) and one week (20% vs 7.8%, p<0.05).28 There was no difference after two weeks postoperatively (3.3% vs 2.2 % at 2 weeks).

Xu et al retrospectively reviewed 1288 patient receiving bipolar enucleation and found that older age and large prostate volume were associated with postoperative stress urinary incontinence. Besides, operation time and blood loss were also reported as risk factors.

Hence many authors used modified methods such as upside down, apical preservation methods, defining the limits of dissection proximal to external sphincter prior to enucleation, in order to reduce postoperative urinary incontinence. Besides pelvic floor exercise was demonstrated to shorten the periods of stress urinary incontinence. However, the role of pelvic floor exercise in enucleation methods in BPH patients are unclear. These questions need further investigations.

6、study aim： To investigate the risk factors of transient incontinence and establish model to predict the incontinence. Besides we will evaluate different surgical methods and treatment methods to improve transient incontinence and the long-term results of different enucleation methods.

7、material and methods： I. study design: prospective cohort study II. . We plan to invite 300 patients whom received enucleation (laser or bipolar) surgery for BPH during 2020 march to 2022 march in National Taiwan University Hospital yun-lin branch to participate this study. We adopted usual care and collect patient's preoperative, intraoperative and postoperative data. The preoperative data include age, comorbidities, medication history, urodynamic parameters and urinary questionnaire. Intraoperative data include operative methods, operative time and surgical complications. Postoperative parameters include urinary questionnaire such as International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF), 4-time use pad questionnaire, IPSS, 7-item Overactive Bladder Symptom Score (OABSS) and urodynamic parameters.

III. Outcome measure

1. Maximum urinary flow rate (Qmax) Prostate volume (TRUSP) , post-voiding residual urine (PVR ) at baseline, 3, 6, 12, and 24-month follow-up visits, pressure-flow study at baseline if indicated.
2. If incontinence and using pad, then biofeedback, ICIQ-SF, 4-item use pad questionnaire every week until incontinence cured. and different type of urinary incontinence such as stress UI, urge UI, total incontinence, mixed incontinence et al
3. IPSS, OABSS instruments, flow, TRUSP and PVR will be scored per instructions for each instrument collected at baseline and at baseline, 3, 6, 12, and 24-month follow-up visits
4. Pre-operative parameters: Age, BMI, comorbidities (DM, Hypertension, heart disease, neurologic disease), anal tone (DRESS), PSA
5. Op parameters: op methods (original en blcok or anterioposterio dissection, preserve 11-1 ocolock) enucleation and morcellation time， catheterization duration,
6. Complication: using modified clavien-dindo classification grade 1-4

ELIGIBILITY:
Inclusion criteria:

* Subject has diagnosis of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction
* Clinical investigator has documented in the subject's medical record that in his/her judgment the subject is a surgical candidate
* Subject is 40 to 90 years of age
* Subject has an IPSS score greater than or equal to 12 measured at the baseline visit
* Subject has medical record documentation of a maximum urinary flow rate (Qmax) less than 15ml/s
* Subject is classified as American Society of Anesthesiologists (ASA) I, II or III

Exclusion criteria:

* Subject has a life expectancy of less than 2 years
* Subject has an active infection (eg, urinary tract infection or prostatitis)
* Subject has a diagnosis of, or has received treatment for, chronic prostatitis or -chronic pelvic pain syndrome (eg, non-bacterial chronic prostatitis)
* Subject has been diagnosed with a urethral stricture or bladder neck contracture
* Subject has history of lower urinary tract surgery (eg, TURP, laser, urinary diversion, artificial urinary sphincter, penile prosthesis)
* Subject has diagnosis of stress urinary incontinence that requires treatment or daily pad/device use
* Subject has diagnosis of prostate cancer and receive cancer treatment
* Subject has a history of carcinoma in situ (CIS), Ta Grade 2, Ta Grade 3 or any T1 stage bladder cancer

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BPH patients need surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-06-02 (Estimated); Study Completion 2024-06-02 (Estimated)

PRIMARY OUTCOMES:
Change of postoperative incontinence from baseline to postoperative 6 months asses by iciq-SF | post-op 1 week, 2 weeks, 3 weeks, 1 month, 2 month, 3 month and 6 months
  change of incontinence severity after operation

SECONDARY OUTCOMES:
Change of postoperative incontinence from baseline to postoperative 6 months asses by 4-item pad questionnaire | post-op 1 week, 2 weeks, 3 weeks, 1 month, 2 month, 3 month and 6 months
  change of pad usage after operation

CONTACTS AND LOCATIONS:
Overall Officials: Shiwei Haung, MDPHD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
need irb approval

REFERENCES:
- [Background] Wei JT, Calhoun E, Jacobsen SJ. Urologic diseases in America project: benign prostatic hyperplasia. J Urol. 2005 Apr;173(4):1256-61. doi: 10.1097/01.ju.0000155709.37840.fe. PMID 15758764
- [Background] Malaeb BS, Yu X, McBean AM, Elliott SP. National trends in surgical therapy for benign prostatic hyperplasia in the United States (2000-2008). Urology. 2012 May;79(5):1111-6. doi: 10.1016/j.urology.2011.11.084. PMID 22546389
- [Background] Reich O, Seitz M, Gratzke C, Schlenker B, Walther S, Stief C. [Benign prostatic hyperplasia (BPH) : Surgical therapy options]. Urologe A. 2010 Jan;49(1):113-26. doi: 10.1007/s00120-009-2183-1. German. PMID 20033128
- [Background] Lourenco T, Pickard R, Vale L, Grant A, Fraser C, MacLennan G, N'Dow J; Benign Prostatic Enlargement team. Minimally invasive treatments for benign prostatic enlargement: systematic review of randomised controlled trials. BMJ. 2008 Oct 9;337:a1662. doi: 10.1136/bmj.a1662. PMID 18845591
- [Background] Reich O, Gratzke C, Bachmann A, Seitz M, Schlenker B, Hermanek P, Lack N, Stief CG; Urology Section of the Bavarian Working Group for Quality Assurance. Morbidity, mortality and early outcome of transurethral resection of the prostate: a prospective multicenter evaluation of 10,654 patients. J Urol. 2008 Jul;180(1):246-9. doi: 10.1016/j.juro.2008.03.058. Epub 2008 May 21. PMID 18499179
- [Background] Issa MM. Technological advances in transurethral resection of the prostate: bipolar versus monopolar TURP. J Endourol. 2008 Aug;22(8):1587-95. doi: 10.1089/end.2008.0192. PMID 18721041
- [Background] Liu JF, Liu CX, Tan ZH, Li SX, Li XZ, Chi N. [Transurethral bipolar plasmakinetic enucleation and resection versus transurethral bipolar plasmakinetic resection of the prostate for BPH: a randomized controlled trial on the incidence of postoperative urinary incontinence]. Zhonghua Nan Ke Xue. 2014 Feb;20(2):165-8. Chinese. PMID 24520671
- [Background] Xu N, Chen SH, Xue XY, Wei Y, Zheng QS, Li XD, Huang JB, Cai H, Sun XL, Lin YZ. Older Age and Larger Prostate Volume Are Associated with Stress Urinary Incontinence after Plasmakinetic Enucleation of the Prostate. Biomed Res Int. 2017;2017:6923290. doi: 10.1155/2017/6923290. Epub 2017 Mar 30. PMID 28466017
- [Background] Nam JK, Kim HW, Lee DH, Han JY, Lee JZ, Park SW. Risk Factors for Transient Urinary Incontinence after Holmium Laser Enucleation of the Prostate. World J Mens Health. 2015 Aug;33(2):88-94. doi: 10.5534/wjmh.2015.33.2.88. Epub 2015 Aug 19. PMID 26331125
- [Background] Goode PS, Burgio KL, Johnson TM 2nd, Clay OJ, Roth DL, Markland AD, Burkhardt JH, Issa MM, Lloyd LK. Behavioral therapy with or without biofeedback and pelvic floor electrical stimulation for persistent postprostatectomy incontinence: a randomized controlled trial. JAMA. 2011 Jan 12;305(2):151-9. doi: 10.1001/jama.2010.1972. PMID 21224456